CLINICAL TRIAL: NCT01616030
Title: Feasibility of Progressive Strength Training in the Early Post Surgical Rehabilitation Period After Hip Fracture Surgery
Brief Title: Early Strength Training After Hip Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Lise Kronborg, Project Physiotherapist, Msc., Copenhagen University Hospital, Hvidovre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH-S-1
Record Dates: First submitted 2012-06-05; First posted 2012-06-11 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Hip Fractures
Keywords: Hip fractures; Strength training
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Strength training, fractured limb (Experimental): Knee-extension strength training of the fractured limb:
  Daily knee-extension strength training with 3 x 10 repetitions using an intensity of 10 Repetition Maximum (RM) for the hip fractured limb started as soon as possible after surgery.
  Interventions: Other: Knee-extension strength training of the fractured limb

INTERVENTIONS:
Other: Knee-extension strength training of the fractured limb — Daily knee-extension strength training with 3 x 10 repetitions using an intensity of 10 Repetition Maximum (RM) for the hip fractured limb started as soon as possible after surgery.

SUMMARY:
Patients treated surgically for a hip fracture have a need of rehabilitation for the regain of former functional skills. Despite an optimized fast track in-hospital rehabilitation program it has been found that patients with hip fracture within 2 weeks after the hip fracture loose more than half of their muscle strength in the fractured limb compared to non-fractured limb. New studies including patients with total hip arthroplasty and strength training applied early after surgery has shown promising results regarding prevention of loss of muscle strength. No similar study has been found including patients with hip fracture.

The purpose of this study is to examine the feasibility of progressive knee-extension strength training of the hip fractured limb, starting Day 1 after surgical treatment for a hip fracture and proceeded every weekday during their hospital stay.

The study will include 20 patients surgically treated for a cervical hip fracture and 20 patients surgically treated for an intertrochanteric or subtrochanteric fracture. All patients are admitted from their own home. Age 60 years or older.

DETAILED DESCRIPTION:
Kronborg L, Bandholm T, Palm H, Kehlet H, Kristensen MT (2014) Feasibility of Progressive Strength Training Implemented in the Acute Ward after Hip Fracture Surgery. PLoS ONE 9(4): e93332. doi:10.1371/journal.pone.0093332

ELIGIBILITY:
Inclusion Criteria:

* Hip fracture diagnosed patients age ≥60 years, admitted to the acute hip fracture unit.
* Medial femoral neck fracture, pertrochanteric fracture or subtrochanteric fracture.
* Ability to speak and understand the Danish language.
* Cognitively well-preserved and able to give personal informed consent no later than by 5th post surgical day.
* Home-residing and with an independent pre-fracture ability to walk equal to New Mobility Score at ≥ 2 indoor.

Exclusion Criteria:

* Multiple fractures
* Postsurgical restrictions of mobilization
* Patient not accepting participation in relevant exercise therapy
* Fracture caused by cancer metastases
* Terminal illness
* Neurological impairment e.g. hemi paresis.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of progression in training loads (kg) during daily knee-extension strength training when commenced immediately after hip fracture surgery. | Baseline to discharge, in average 10 days.
  Feasibility is evaluated on the basis of adherence to program, adverse events, target training intensity, hip pain during training and other potential restricting factors, e.g. confusion, exhaustion and dropouts.

SECONDARY OUTCOMES:
Change in maximum isometric knee-extension strength and strength deficits, fractured % of non-fractured limb measured by handheld dynamometer. | Baseline to discharge, in average 10 days.

OTHER OUTCOMES:
Association between 10 meter fast speed walk and knee-extension strength discharge from hospital. | Day before discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, PhD, Study Director — Copenhagen University Hospital at Hvidovre, Denmark
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Result] Kronborg L, Bandholm T, Palm H, Kehlet H, Kristensen MT. Feasibility of progressive strength training implemented in the acute ward after hip fracture surgery. PLoS One. 2014 Apr 3;9(4):e93332. doi: 10.1371/journal.pone.0093332. eCollection 2014. PMID 24699276